CLINICAL TRIAL: NCT05851573
Title: Stepped Care Model of Psychological Care for Aphasia
Brief Title: Stepped Care for Aphasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Deena Blackett, Principal Investigator, Medical University of South Carolina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00125313
Record Dates: First submitted 2023-04-07; First posted 2023-05-09 (Actual); Results first posted 2025-02-24 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Aphasia; Stroke
MeSH Terms: conditions — Aphasia; Stroke | interventions — Psychosocial Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Psychosocial intervention (Experimental)
  Interventions: Behavioral: Psychosocial intervention

INTERVENTIONS:
Behavioral: Psychosocial intervention — an SLP-administered 5-week treatment focused on psychological well-being

SUMMARY:
This study is recruiting people who had a stroke at least 1 month ago and now have a language impairment called aphasia. Living with aphasia can have devastating effects on communication and quality of life, and it is not uncommon for survivors with aphasia to face psychological problems like depression and anxiety. Participants who are eligible for this study will undergo baseline testing, engage in a 5-week treatment focused on psychological well-being, undergo post-treatment testing, and then testing again 1-month later. Check-in phone calls will be conducted during the 1-month off period and participants will be interviewed about their experience at the end of the study as well. Compensation will be provided to participants with aphasia.

ELIGIBILITY:
Inclusion Criteria:

* 18-81 years old
* Native English speaker (English fluency by age 7)
* Aphasia as a result of a left-hemisphere ischemic or hemorrhagic stroke (WAB-R Aphasia Quotient < 93.8)
* At least 1-month post-stroke
* Confirmation of left hemisphere stroke per medical records
* Discharged from hospital
* Participant is willing and able to consent for themselves.

Exclusion Criteria:

* Uncorrected hearing or visual impairment that prevents completion of experimental activities as determined by self-report
* History of other neurological disorder or disease beside stroke (e.g., dementia, traumatic brain injury) as determined by self-report and/or medical records
* Self-reported history of premorbid learning disability
* Severe auditory comprehension deficits (as indicated by a score of more than two standard deviations below norms on the Auditory Verbal section of WAB-R)

Ages: 18 Years to 81 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2023-03-31 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Interested participants provided informed consent and were then screened to determine if they meet all eligibility criteria. After enrollment, all participants were assigned to the same intervention arm.
Period: Overall Study
Arm/Group | Psychosocial Intervention
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Psychosocial Intervention
Number analyzed (Participants) | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.6 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 11
Western Aphasia Battery-Revised Aphasia Quotient [Mean (Standard Deviation); unit: units on a scale] — Western Aphasia Battery - Revised Aphasia Quotient: This is a measure of overall aphasia severity (severity of language impairment) and is calculated based on performance on the subscales included on the WAB-R per WAB-R scoring protocols. The total range of this scale is 0 to 100. A higher score indicates better language function (less severe aphasia).
  units on a scale | 74.0 (18.0)
Months Post-Stroke [Mean (Standard Deviation); unit: months] | 43.6 (41.1)
Years of Education [Mean (Standard Deviation); unit: years] | 15.8 (2.9)
Cognitive Assessment of Stroke Patients [Mean (Standard Deviation); unit: units on a scale] — The Cognitive Assessment of Stroke Patients is a measure of general cognitive function for stroke survivors. The total range of this measure is 0 to 36. Higher scores indicate better cognitive function.
  units on a scale | 30.3 (2.5)

OUTCOME MEASURES:

1. Primary Outcome: Change in the Depression Score on Hospital Anxiety and Depression Scale at Post-Intervention
Description: Change in the total depression Hospital Anxiety and Depression Scale scores between baseline and post-treatment (baseline-post-treatment). Minimum score 0, maximum score 21. Positive scores indicate an improvement in symptoms, negative scores indicate a worsening in symptoms.
Time Frame: through intervention completion, an average of 7 weeks
Population: One participant was excluded due to missing HADS data at post-intervention.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Psychosocial Intervention
Number analyzed (Participants) | 10
units on a scale | 2.2 (2.82)
Statistical Analysis 1: Comparison: Psychosocial Intervention; Test type: Other; p < .05, t-test, 2 sided; df = 9

2. Primary Outcome: Change in the Anxiety Score on Hospital Anxiety and Depression Scale at Post-Intervention
Description: Change in the total anxiety Hospital Anxiety and Depression Scale scores between baseline and post-treatment (baseline-post-treatment). Minimum score 0, maximum score 21. Positive scores indicate an improvement in symptoms, negative scores indicate a worsening in symptoms.
Time Frame: through intervention completion, an average of 7 weeks
Population: One participant was excluded due to missing HADS data at post-intervention.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Psychosocial Intervention
Number analyzed (Participants) | 10
units on a scale | 0.40 (4.30)
Statistical Analysis 1: Comparison: Psychosocial Intervention; Test type: Other; p = .775, t-test, 2 sided; df = 9

3. Secondary Outcome: Change in Dynamic Visual Analogue Mood Scales at Post-Intervention
Description: Total summary score (min: 0, max: 100, higher scores indicate better outcome) and sadness score (min: 0, max: 100, higher scores indicate better outcome) (baseline-post-treatment). Positive number indicate worsening in mood, negative numbers indicate an improvement in mood.
Time Frame: through study completion, an average of 7 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Psychosocial Intervention
Number analyzed (Participants) | 11
units on a scale | -4.18 (17.42)
Statistical Analysis 1: Comparison: Psychosocial Intervention; Test type: Other; p = .444, t-test, 2 sided; df = 10

4. Secondary Outcome: Change in Stroke Aphasia Depression Questionnaire - 10 at Post-Intervention
Description: Total score (min: 0, max: 30, higher scores indicate worse outcome); baseline-post-treatment; positive scores indicate improvement in symptoms, negative score indicate worsening of symptoms
Time Frame: through intervention completion, an average of 7 weeks
Population: One participant was missing data on SADQ-10 at post-intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Psychosocial Intervention
Number analyzed (Participants) | 10
units on a scale | 0.10 (5.9)
Statistical Analysis 1: Comparison: Psychosocial Intervention; Test type: Other; p = .959, t-test, 2 sided; df = 9

5. Secondary Outcome: Change in Behavioural Outcomes of Anxiety Scale at Post-Intervention
Description: Total score (min: 0, max: 30, higher scores indicate worse outcome); baseline-post-intervention; positive scores indicate an improvement in symptoms, negative scores indicate a worsening in symptoms.
Time Frame: through intervention completion, an average of 7 weeks
Population: One participant was missing data from this measure at baseline.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Psychosocial Intervention
Number analyzed (Participants) | 10
units on a scale | 2.00 (3.01)
Statistical Analysis 1: Comparison: Psychosocial Intervention; Test type: Other; p = .068, t-test, 2 sided; df = 9

6. Secondary Outcome: Change in Modified Perceived Stress Scale at Post-Intervention
Description: Total score (min: 0, max: 40, higher scores indicate worse outcome); baseline-post-intervention; positive numbers indicate an improvement in symptoms, negative numbers indicate a worsening in symptoms
Time Frame: through intervention completion, an average of 7 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Psychosocial Intervention
Number analyzed (Participants) | 11
units on a scale | 3.36 (6.55)
Statistical Analysis 1: Comparison: Psychosocial Intervention; Test type: Other; p = .119, t-test, 2 sided; df = 10

7. Secondary Outcome: Change in Stroke Aphasia Quality of Life - 39 at Post-Intervention
Description: Total score (min: 1, max: 5), baseline-post-intervention, positive numbers indicate a worsening of quality of life, negative numbers indicate an improvement in quality of life
Time Frame: through intervention completion, an average of 7 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Psychosocial Intervention
Number analyzed (Participants) | 11
units on a scale | -.093 (.258)
Statistical Analysis 1: Comparison: Psychosocial Intervention; Test type: Other; p = .258, t-test, 2 sided; df = 10

8. Secondary Outcome: Change in Communication Confidence Rating Scale for Aphasia at Post-Intervention
Description: Total score (min: 10, max: 40, higher scores indicate better confidence); baseline-post-intervention, positive numbers indicate a worsening in communication confidence and negative numbers indicate an improvement in communication confidence
Time Frame: through intervention completion, an average of 7 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Psychosocial Intervention
Number analyzed (Participants) | 11
units on a scale | -.818 (4.92)
Statistical Analysis 1: Comparison: Psychosocial Intervention; Test type: Other; p = .593, t-test, 2 sided; df = 10

ADVERSE EVENTS:
Time Frame: up to 11 weeks
Description: Participants were monitored for adverse events for the duration that the participant was enrolled from their baseline session to their 1-month follow-up session, which, for most participants, was about 11 weeks.
Arm/Group | Psychosocial Intervention
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-12-17): https://cdn.clinicaltrials.gov/large-docs/73/NCT05851573/Prot_SAP_001.pdf
  • Informed Consent Form (2023-02-23): https://cdn.clinicaltrials.gov/large-docs/73/NCT05851573/ICF_000.pdf